CLINICAL TRIAL: NCT00000730
Title: A Randomized, Comparative Trial of Trimetrexate With Leucovorin Rescue Versus Standard Anti-Pneumocystis Therapy Versus Standard Anti-Pneumocystis Therapy With High Dose Steroids for AIDS Patients With Pneumocystis Pneumonia Who Appear to Be Refractory to Conventional Drugs
Brief Title: Comparison of Three Treatments for Pneumocystis Pneumonia in AIDS Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: ACTG 030; 11006 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; Trimetrexate; AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Leucovorin; Folic Acid Antagonists; Acquired Immunodeficiency Syndrome; Antiprotozoal Agents; Sulfamethoxazole-Trimethoprim
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — trimetrexate glucuronate; Methylprednisolone; Pentamidine; Trimethoprim, Sulfamethoxazole Drug Combination; Leucovorin

INTERVENTIONS:
Drug: Trimetrexate glucuronate
Drug: Methylprednisolone
Drug: Pentamidine isethionate
Drug: Sulfamethoxazole-Trimethoprim
Drug: Leucovorin calcium

SUMMARY:
This study compares three different therapies for treatment of refractory Pneumocystis carinii pneumonia (PCP) in patients with AIDS. "Refractory" means that the patient has failed to respond to at least 4 days of treatment with either of two standard therapies: (1) sulfamethoxazole/trimethoprim (SMX/TMP) or (2) pentamidine (PEN). This study compares therapy with trimetrexate (TMTX) and leucovorin (LCV) to standard therapy and standard therapy plus high-dose steroids (methylprednisolone). The purpose is to find better and safer forms of treatment for PCP in AIDS patients. There is at present no scientific information about the best treatment for an AIDS patient with PCP who is not improving while receiving the standard therapies (SMX/TMP or PEN). New drug treatments are available, including steroid therapy and TMTX, but there is no information proving that these new treatments work better than the standard therapies.

DETAILED DESCRIPTION:
There is at present no scientific information about the best treatment for an AIDS patient with PCP who is not improving while receiving the standard therapies (SMX/TMP or PEN). New drug treatments are available, including steroid therapy and TMTX, but there is no information proving that these new treatments work better than the standard therapies.

Hospitalized patients who have failed to respond to at least 4 full days but no greater than 14 full days of therapy with SMX/TMP or PEN are randomly placed into one of three study groups. Patients are stratified for (1) mechanical ventilation at enrollment, (2) prior zidovudine therapy of at least 4 weeks duration, and (3) first versus subsequent episode of PCP. One group of patients receives TMTX by intravenous infusion for 21 days and LCV for 24 days. The second and third group of patients receive either PEN or SMX/TMP depending on which therapy they have already received and not improved on. The difference between the second and third group is that the second group receives the conventional therapy (PEN or SMX/TMP) and a placebo (inactive medication) and the third group receives the conventional therapy and prednisolone. Neither investigators nor patients know whether patients receive methylprednisolone. Patients continue study treatment until a study end point is reached or for a minimum of 21 days (unless there is toxicity).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* physiologic replacement doses of steroids.
* Pneumocystis carinii pneumonia (PCP) in patient who is HIV positive by ELISA, HIV culture, or p24 antigenemia, or is a member of a risk group for HIV infection.
* Failed at least 4 but not > 14 full days' therapy with either sulfamethoxazole/trimethoprim (SMX/TMP) or parenteral pentamidine. Patients must have received therapy with only one of the two conventional agents prior to enrollment.
* Patients in whom an unequivocal diagnosis of this episode of PCP has been or can be established by morphologic confirmation of three or more typical Pneumocystis carinii organisms in sputum, bronchoalveolar lavage fluid, or lung tissue obtained by transbronchial or open lung biopsy within 15 days prior to study entry.
* Patients in whom no significant improvement in arterial-alveolar oxygen pressure (defined as a decrease of at least 15mm Hg) is observed in the 24 hours prior to entry.
* Patient is willing to have maximal medical support, including pressors, invasive monitoring, and/or mechanical ventilation, during at least the first 7 days of protocol therapy if such support is necessary. Continuation of maximal medical support beyond 7 days is at discretion of investigator and patient.
* Patients with history of hypersensitivity less severe than type I may be enrolled if, in opinion of investigator, these adverse effects do not prohibit rechallenge with the drug.

Prior Medication:

Required:

* At least 4 full days but no greater than 14 full days of parenteral and/or oral therapy with sulfamethoxazole/trimethoprim (SMX/TMP) or pentamidine.

Allowed:

* Zidovudine (AZT).

Exclusion Criteria

Co-existing Condition:

Excluded:

* Patients with history of type I hypersensitivity (urticaria, angioedema, anaphylaxis), exfoliative dermatitis, or other life-threatening reaction secondary to trimetrexate, sulfamethoxazole/trimethoprim, or pentamidine.
* Presence of any process that, in the opinion of investigator, would be adversely and seriously affected by steroid therapy.
* Failure to meet inclusion criteria.

Concurrent Medication:

Excluded:

* Zidovudine (AZT).
* Myelosuppressive agents.
* Nephrotoxic agents.
* AZT may be resumed at completion of study.

Excluded:

* Patients with history of type I hypersensitivity (urticaria, angioedema, anaphylaxis), exfoliative dermatitis, or other life-threatening reaction secondary to trimetrexate, sulfamethoxazole/trimethoprim, or pentamidine.
* Presence of any process that, in the opinion of investigator, would be adversely and seriously affected by steroid therapy.
* Failure to meet inclusion criteria.

Prior Medication:

Excluded within 4 days of study entry:

* Any other investigational agent.
* Excluded within 14 days of study entry:
* Steroids (other than physiologic replacement doses).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240
Dates: Study Completion 1989-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masur H, Study Chair
Locations (1):
- Julio Arroyo, West Columbia, South Carolina, United States

REFERENCES:
- [Background] Amsden GW, Kowalsky SF, Morse GD. Trimetrexate for Pneumocystis carinii pneumonia in patients with AIDS. Ann Pharmacother. 1992 Feb;26(2):218-26. doi: 10.1177/106002809202600217. PMID 1532518